CLINICAL TRIAL: NCT05244070
Title: A Phase 1, Multicenter, Open-label Study of BMS-986403 in Subjects With Relapsed and/or Refractory Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL)
Brief Title: A Study to Evaluate the Safety and Tolerability of BMS-986403 in Participants With Relapsed and/or Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA097-001; 2021-003274-31 (EudraCT Number)
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma
Keywords: BMS-986403; Relapsed and/or Refractory; Small Lymphocytic Lymphoma (CLL); Chronic Lymphocytic Leukemia (SLL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BMS-986403 + Fludarabine + Cyclophosphamide (Experimental)
  Interventions: Drug: BMS-986403; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: BMS-986403 — Specified dose on specified days
Drug: Fludarabine — Specified dose on specified days
Drug: Cyclophosphamide — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the safety and preliminary efficacy of BMS-986403 in participants with relapsed and/or refractory chronic lymphocytic leukemia (R/R CLL) or small lymphocytic lymphoma (SLL).

ELIGIBILITY:
Inclusion Criteria:

* Participants with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) and high-risk features must have failed at least 2 lines of prior therapy and participants with CLL or SLL and standard risk features must have failed at least 3 lines of prior therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
* Either currently has central vascular access or is a candidate to receive central vascular access or peripheral vascular access for leukapheresis procedure
* Has recovery to Grade ≤ 1 or baseline of any non-hematologic toxicities due to previous therapy, except alopecia (any Grade acceptable) and peripheral neuropathy (Grade ≤ 2 acceptable)

Exclusion Criteria:

* Any condition, including active or uncontrolled infection, or the presence of laboratory abnormalities, that places the subject at unacceptable risk if they were to participate in the study
* Systemic fungal, bacterial, viral, or other infection that is not controlled
* Active autoimmune disease requiring immunosuppressive therapy
* Progressive deep vein thrombosis or pulmonary embolism requiring treatment, but not yet on a stable anticoagulation regimen

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 2 years after BMS-986403 infusion
Number of participants with serious adverse events (SAEs) | Up to 2 years after BMS-986403 infusion
Number of participants with clinical laboratory abnormalities | Up to 2 years after BMS-986403 infusion
Number of participants with dose-limiting toxicity (DLT) | Up to 2 years after BMS-986403 infusion
Maximum-tolerated dose (MTD) based on the incidence of DLTs that occur during the DLT evaluation period | Up to 2 years after BMS-986403 infusion
Recommended Phase 2 Dose (RP2D) based on the incidence of DLTs that occur during the DLT evaluation period | Up to 2 years after BMS-986403 infusion

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years after BMS-986403 infusion
Complete remission rate (CRR) | Up to 2 years after BMS-986403 infusion
Duration of response (DOR) | Up to 2 years after BMS-986403 infusion
Duration of complete remission (DOCR) | Up to 2 years after BMS-986403 infusion
Time to response (TTR) | Up to 2 years after BMS-986403 infusion
Time to CR (TTCR) | Up to 2 years after BMS-986403 infusion
Progression free survival (PFS) | Up to 2 years after BMS-986403 infusion
Overall survival (OS) | Up to 2 years after BMS-986403 infusion
Pharmacokinetics by polymerase chain reaction (PCR): Maximum concentration (Cmax) | Up to 2 years after BMS-986403 infusion
Pharmacokinetics by PCR: Time to peak (maximum) concentration (Tmax) | Up to 2 years after BMS-986403 infusion
Pharmacokinetics by PCR: Area under the curve (AUC) | Up to 2 years after BMS-986403 infusion

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (9):
- United States (6):
  - Local Institution - 0005, Birmingham, Alabama
  - Local Institution - 0016, Duarte, California
  - Local Institution - 0007, Boston, Massachusetts
  - Local Institution - 0026, Hackensack, New Jersey
  - Local Institution - 0009, Columbus, Ohio
  - Local Institution - 0002, Seattle, Washington
- Spain (3):
  - Local Institution - 0024, Barcelona
  - Local Institution, Madrid
  - Local Institution, Salamanca

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com